CLINICAL TRIAL: NCT03981939
Title: Perianal Fistula Procedure Validation, Matched Case Control, and Patient Journey Study
Brief Title: Perianal Fistula (PAF) Validation and Burden of Illness Study
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5009; U1111-1233-6312 (Other: World health organization)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Disease; Perianal Fistula; Crohns Disease
Keywords: Drug therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CD Participants with CPAF - The Ottawa Hospital (TOH): Participants diagnosed with Complex Perianal Fistula (CPAF) from the Ottawa Hospital (TOH) were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
  Interventions: Other: No intervention
- CD Participants without CPAF (ICES database): Participants diagnosed with CD and without CPAF from Institute for Clinical Evaluative Sciences (ICES) database who did not meet the case definition were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
  Interventions: Other: No intervention
- CD Participants with CPAF (ICES database): Participants with CD and CPAF from ICES database who met the case definition were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, participants did not receive any intervention in this study and were only observed retrospectively.

SUMMARY:
The purpose of this study is to gain a better understanding of the disease burden and unmet need of perianal fistulas within Crohn's disease (CD) in Ontario.

DETAILED DESCRIPTION:
This is a retrospective follow-up observational study of participants with CD with and without complex perianal fistula (CPAF) from January 2002 to March 2017. The study will verify the potential of using procedure codes to reliably identify participants with CPAF in Validation Study (Objective 1), compare Crohn's participants with CPAF (cases) to matched participants without CPAF (controls) to determine the disease burden and healthcare resource utilization of Crohn's related CPAF in Ontario, and will describe the participant's journey among Crohn's participants following the first diagnosis of CPAF (Objective 3).

The study will enroll approximately 600 participants (300 participants with CPAF and 300 participants without CPAF). All participants will be enrolled in 2 observation groups:

* CD Participants with/without CPAF (ICES data)
* CD Participants with CPAF - The Ottawa Hospital (TOH)

The data will be collected through Ontario health administrative data. Participants will be observed retrospectively who were diagnosed with CD with and without fistula between index period: April 2002 and July 2013. Participants will be followed up retrospectively from the index period (that is onset of CPAF) to the end of study (Objective 2), and for 5 years following the (Objective 3) index date defined as onset of CPAF will be selected based on the first time they meet the first code in the case definition identified in Objective 1 between April 1, 2005 to March 31, 2012. The overall time for data collection in this study will be approximately 7 months.

ELIGIBILITY:
Inclusion Criteria for Objective 1:

1. Inclusion in the TOH "reference" database.
2. Aged 18-105 inclusive at date of index.
3. Participant can be linked between TOH "reference" database to the Institute for Clinical Evaluative Sciences (ICES) databases based on health card number.
4. Incident inclusion in the Ontario Crohn's and Colitis Cohort (OCCC) between April 1, 2002 to July 1, 2013.
5. Incident diagnosis of CPAF in TOH database between April 1, 2004 to July 1, 2015.

Inclusion Criteria for Objective 2:

1. Participants were incident in the OCCC from April 1, 2002 to March 31, 2012.
2. The case meets the PAF case definition identified in Objective 1 in the selection period (April 1, 2005 to March 31, 2012).
3. Aged 18-105 inclusive at date of index.

Inclusion Criteria for Objective 3:

1. Inclusion in the OCCC at or prior to index visit with a diagnosis of Crohn's disease.
2. The case meets the CPAF case definition identified in Objective 1 in the selection period.
3. Have to have 5 years of follow-up.
4. Aged 18-105 inclusive at date of index.

Exclusion Criteria for Objective 1:

1. Missing demographics at index date (sex, age, Local Health Integration Network (LHIN), income quintile) in all databases.
2. Death date in the ICES data prior to TOH CPAF incidence date.

Exclusion Criteria for Objective 2:

1. Missing demographics at index date (sex, age, neighbourhood income quintile, LHIN).
2. Death during 5-year analysis period.
3. Ontario Health Insurance Plan (OHIP) coverage is terminated during the follow-up example if the participant moves to another province.
4. Meeting the case definition during the lookback period.
5. Cases for whom a matched control cannot be found.

Exclusion Criteria for Objective 3:

1. Missing demographics at index date (sex, age, neighbourhood income quintile, LHIN).
2. Death during 5-year analysis period.
3. OHIP coverage is terminated during the 5-year analysis period example if the participant moves to another province.
4. Meeting the case definition during the lookback period.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CD with and without CPAF will be observed retrospectively in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3032 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical director, Study Director — Takeda
Locations (1):
- Takeda Canada, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from participants were collected for this retrospective observational study at a single investigative site in Canada from 2 July 2019 to 31 December 2019.
Pre-assignment Details: Participants with a diagnosis of Crohn's disease (CD) with and without Complex Perianal Fistula (CPAF) were enrolled from The Ottawa Hospital (TOH) and Institute for Clinical Evaluative Sciences (ICES) database and were observed retrospectively in this study.
Groups:
- CD Participants With CPAF - The Ottawa Hospital (TOH): Participants diagnosed with CPAF from TOH were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
- CD Participants Without CPAF (ICES Database): Participants diagnosed with CD and without CPAF from ICES database who did not meet the case definition were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
Period: Overall Study
Arm/Group | CD Participants With CPAF - The Ottawa Hospital (TOH) | CD Participants Without CPAF (ICES Database) | CD Participants With CPAF (ICES Database)
Started | 549 | 1902 | 581
Completed | 549 | 1902 | 581
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants with CD, with CPAF or without CPAF from TOH and ICES database were included in the analysis.
Groups:
- CD Participants With CPAF - TOH: Participants diagnosed with CPAF from TOH were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
- Total: Total of all reporting groups
Arm/Group | CD Participants With CPAF - TOH | CD Participants Without CPAF (ICES Database) | CD Participants With CPAF (ICES Database) | Total
Number analyzed (Participants) | 549 | 1902 | 581 | 3032
Age, Continuous [Mean (Full Range); unit: years] | 38.12 [26.3 to 48] | 31.83 [23 to 38] | 33.09 [23 to 40] | 34.34 [23 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 903 | 279 | 1486
  Male | 245 | 999 | 302 | 1546
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 549 | 1902 | 581 | 3032

OUTCOME MEASURES:

1. Primary Outcome: Objective 1: Number of CD Participants Who Have CPAF Using Various Codes in an TOH Database
Description: Index date first time participant meets case definition(diagnosis of CD with CPAF in index period).Participants divided as:2 diagnosis/imaging codes(IC),2 codes must be in 2 year(yr) period of each other;3 diagnosis/IC/intervention code/EUA+seton;3 diagnosis/IC/intervention code/EUA+seton,diagnosis/IC requirements are satisfied,codes must be in 2yr period of each other;2 diagnosis/IC;3 diagnosis/IC,3 codes must be in 2yr period of each other;3 diagnosis/IC;diagnosis/IC+(EUA+Seton);diagnosis/IC+(EUA+Seton),2 codes must be in 2yr period of each other;3 diagnosis /IC+intervention code 4 codes must be in 2 yr period of each other;2 IC/intervention code/diagnosis code/EUA+seton;2 IC/intervention code/diagnosis code/EUA+seton,IC requirements are satisfied, codes must be in 2yr period of each other;2 diagnosis/IC+intervention code;3 diagnosis/IC+intervention code;2 diagnosis/IC+intervention code,3 codes must be in 2yr period of each other;diagnosis/imaging/intervention codes;diagnosis/IC.
Time Frame: From the date of CD diagnosis up to the index date (approximately 5 years)
Population: All participants identified from TOH with and without CPAF were included in the analysis. Participants could meet more than more case definition.
Measure: Count of Participants; unit: Participants
Arm/Group | CD Participants With CPAF - TOH
Number analyzed (Participants) | 549
Participants
  Any 2 Diagnosis/IC, in a 2 Year Period of Each Other | 120
  Any 3 Diagnosis/ IC/ Intervention Code/EUA+seton | 120
  Any 3 Diagnosis/ IC/ Intervention/EUA+seton, Diagnosis/ IC Requirements are Satisfied | 127
  Any 2 Diagnosis/ IC | 127
  Any 3 Diagnosis/ IC, 3 Codes Must be in 2 Year Period of Each Other | 88
  Any 3 Diagnosis/ IC | 97
  Any Diagnosis/ IC + (EUA+ Seton) | 83
  Any Diagnosis/ IC + (EUA+Seton), in a 2 Year Period of Each Other | 78
  Any 3 Diagnosis/IC + Intervention Code, 4 Codes Must be in 2 Year Period of Each Other | 66
  Any 2 IC Intervention Code/ Diagnosis Code/EUA+Seton | 127
  Any 2 Imaging/Intervention/ Diagnosis Code/EUA+seton, If Imaging Code Requirements Are Satisfied | 127
  Any 2 Diagnosis/ IC + Intervention Code | 69
  Any 3 Diagnosis/ IC + an Intervention Code | 67
  Any 2 Diagnosis/ IC + Intervention Code, 3 Codes Must be in 2 Year Period of Each Other | 69
  Any Diagnosis/ IC / Intervention Codes | 146
  Any Diagnosis/ IC | 146

2. Primary Outcome: Objective 2: Mean Costs for Crohn's Disease Participants With and Without CPAF in ICES Database CPAF
Description: Impact of total disease burden on participants CD with and without CPAF was measured as total cost and cost by sector which included general physicians (GP), specialist, all physician OHIP, home care services, hospital admissions, dialysis, cancer, and radiation, emergency department (ED), Ontario drug benefit (ODB), hospital outpatient clinics, same day surgery (SDS). Index date was defined as the date the first time the participant meets the case definition i.e. diagnosis of CD with CPAF in the index period.
Time Frame: From the index date up to end of study (approximately 5 years post-index)
Population: All participants who were eligible as cases (CD Participants with CPAF) and controls (CD Participants without CPAF) from the ICES database were used in the analysis.
Measure: Mean (Standard Deviation); unit: canadian dollars
Arm/Group | CD Participants Without CPAF (ICES Database) | CD Participants With CPAF (ICES Database)
Number analyzed (Participants) | 1902 | 581
canadian dollars
  Total Cost | 32781.12 (52124.77) | 62375.54 (70332.9)
  Total Cost (Without ODB) | 22866.85 (37256.27) | 36486.07 (42218.43)
  Cost by Sector: General Physicians (GP) | 1192.63 (2936.3) | 1275.58 (1974.01)
  Cost by Sector: Specialist | 5978.09 (5317.74) | 8075.60 (5777.89)
  Cost by Sector: All physician OHIP | 8029.55 (6818.29) | 10368.04 (6969.59)
  Cost by Sector: Home Care Services | 900.90 (14925.27) | 4142.01 (12246.05)
  Cost by Sector: Hospital Admissions | 7586.89 (23760.92) | 11079.55 (24994.66)
  Cost by Sector: Dialysis, Cancer, and Radiation | 64.61 (949.45) | 275.93 (4181.82)
  Cost by Sector: Non-hospital Based Residential Care | 182.73 (2797.46) | 217.79 (2781.88)
  Cost by Sector: Emergency Department (ED) | 1421.81 (2167.73) | 1807.10 (2658.28)
  Cost by Sector: ODB | 9917.46 (32562.86) | 25889.50 (52074.97)
  Cost by Sector: Hospital Outpatient Clinics | 3177.37 (3632.82) | 5660.54 (5234.69)
  Cost by Sector: Same Day Surgery (SDS) | 1500.39 (1504.51) | 2935.31 (2270.25)

3. Primary Outcome: Objective 2: Number of Visits for Healthcare Resource Utilization for Crohn's Disease Participants With and Without CPAF in ICES Database
Description: Healthcare Resource Utilization was based on three procedures which included the number of ED visits, number of hospitalizations and number of outpatient visits. Index date was defined as the date the first time the participant meets the case definition i.e. diagnosis of CD with CPAF in the index period.
Time Frame: From the index date up to end of study (approximately 5 years post-index)
Population: All participants who were eligible as cases (CD Participants with CPAF) and controls (CD Participants without CPAF) from the ICES database were included in the analysis.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | CD Participants Without CPAF (ICES Database) | CD Participants With CPAF (ICES Database)
Number analyzed (Participants) | 1902 | 581
visits
  Number of ED Visits | 4.26 (6.28) | 5.57 (8.09)
  Number of Hospitalizations | 0.95 (1.74) | 1.38 (2.00)
  Number of Outpatient Visits | 8.57 (9.81) | 15.18 (14.07)

4. Primary Outcome: Objective 3: Mean Costs Based on Three Procedures for Crohn's Disease Participants With CPAF by Sector in ICES Database
Description: Impact of total disease burden on participants CD with CPAF was based on three procedures which included total cost, total cost (without ODB) and cost by sector i.e. general physicians (GP), specialist, all physician OHIP, home care services, hospital admissions, Dialysis, Cancer, and Radiation, non-hospital based residential care, emergency department (ED), Ontario drug benefit (ODB), hospital outpatient clinics, same day surgery (SDS). Index date was defined as the date the first time the participant meets the case definition i.e. diagnosis of CD with CPAF in the index period. Participants with CD and CPAF were categorized into pre-defined treatment pathways and results are reported in three arms: No Intervention, EUA ± Seton and Advanced Intervention.
Time Frame: From the index date up to 5 years post-index
Population: All participants who were eligible as cases (CD Participants with CPAF) CPAF from the ICES database were included in the analysis.
Measure: Mean (Standard Deviation); unit: canadian dollars
Groups:
- No Intervention: Participants with CD and CPAF who did not receive any interventions following their first diagnosis of CPAF and were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
- Exam Under Anesthesia (EUA) ± Seton Only: Participants with CD and CPAF received only EUA ± seton as part of their treatment, with no additional procedures administered in this group and were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
- Advanced Intervention: Participants with CD and CPAF received 2 x EUA ± seton and single EUA ± seton, followed by an advanced intervention or diversion procedure. The participants who did not receive EUA ± seton received advanced intervention or diversion as their 1st line of treatment in this group and were observed retrospectively in this arm group for the index period (April 1, 2007 to March 31, 2013).
Arm/Group | No Intervention | Exam Under Anesthesia (EUA) ± Seton Only | Advanced Intervention
Number analyzed (Participants) | 237 | 307 | 37
canadian dollars
  Total Cost | 45982.45 (51581.52) | 65430.16 (68268.35) | 142034.86 (119455.5)
  Total Cost (Without ODB) | 26799.65 (26777.44) | 36992.93 (33981.36) | 94326 (100709.22)
  Cost by Sector: GP | 1144.88 (1762.59) | 1218.24 (1583.95) | 2588.51 (4379.07)
  Cost by Sector: Specialist | 7128.15 (5772.59) | 8019.46 (4884.16) | 14610.30 (8173.77)
  Cost by Sector: All physician OHIP | 9293.98 (6771.63) | 10240.95 (5951.3) | 18302.27 (10416.85)
  Cost by Sector: Home Care Services | 1231.69 (3596.56) | 5217.44 (14078.41) | 13860.7 (21997.79)
  Cost by Sector: Hospital Admissions | 7615.50 (14938.04) | 9623.01 (18429.69) | 45353.59 (66413.97)
  Cost by Sector: Dialysis, Cancer, and Radiation | 212.03 (2312.88) | 350.46 (5383.99) | 66.78 (406.23)
  Cost by Sector: Non-Hospital Based Residential Care | 293.11 (3402.11) | 185.89 (2393.87) | 0.00 (0.00)
  Cost by Sector: Emergency department (ED) | 1664.22 (2355.68) | 1657.65 (1966.21) | 3962.38 (6285.67)
  Cost by Sector: ODB | 19182.85 (42673.84) | 28437.24 (55455.37) | 47708.86 (69074.61)
  Cost by Sector: Hospital Outpatient Clinics | 4482.35 (4128.71) | 6202.11 (5617.27) | 8713.70 (6348.41)
  Cost by Sector: SDS | 2007.24 (2090.86) | 3515.43 (2132.19) | 4066.57 (2424.82)

5. Primary Outcome: Objective 3: Number of Visits for Healthcare Resource Utilization Based on Three Procedures for Crohn's Disease Participants With CPAF
Description: Healthcare Resource Utilization was based on three procedures which included the number of ED visits, number of hospitalizations and number of outpatient visits. Index date was defined as the date the first time the participant meets the case definition i.e. diagnosis of CD with CPAF in the index period. Participants with CD and CPAF were categorized into pre-defined treatment pathways and results are reported in three arms: No Intervention, EUA ± Seton and Advanced Intervention.
Time Frame: From the index date up to 5 years post-index
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | No Intervention | Exam Under Anesthesia (EUA) ± Seton Only | Advanced Intervention
Number analyzed (Participants) | 237 | 307 | 37
visits
  Number of ED Visits | 5.29 (7.74) | 5.11 (5.79) | 11.22 (18.46)
  Number of Hospitalizations | 1.06 (1.54) | 1.37 (1.84) | 3.57 (3.79)
  Number of Outpatient Visits | 12.11 (11.31) | 16.57 (15.04) | 23.24 (16.82)

ADVERSE EVENTS:
Time Frame: Approximately 5 years
Description: Data of adverse events or adverse drug reactions were not collected as part of the study database.
Arm/Group | CD Participants With CPAF - The Ottawa Hospital (TOH) | CD Participants Without CPAF (ICES Database) | CD Participants With CPAF (ICES Database)
All-Cause Mortality (participants affected / at risk) | 0/549 | 0/1902 | 0/581
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03981939/Prot_SAP_000.pdf